CLINICAL TRIAL: NCT01354951
Title: Phase II Study Assessing the Potential for Reduced Toxicity Using Focal Brachytherapy Early Stage, Low Volume in Prostate Cancer
Brief Title: Assessing the Potential for Reduced Toxicity Using Focal Brachytherapy in Early Stage, Low Volume Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Colorado, Denver (Other); M.D. Anderson Cancer Center (Other); Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-056
Record Dates: First submitted 2011-05-16; First posted 2011-05-17 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2017-11

CONDITIONS: Prostate Cancer
Keywords: Focal Brachytherapy; Endorectal coil MRI; Quality of Life; 11-056
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (1):
- Prostate Biopsy, Focal Brachytherapy , Assessment of QOL (Experimental): This is a non-randomized, Phase II study examining the tolerance profile (primary endpoint) as well as the secondary endpoints of QOL changes, efficacy and the correlation of post-treatment MRI findings with post-treatment biopsy outcomes in men with early stage low volume prostate cancer treated with focal brachytherapy.
  Interventions: Other: Prostate Biopsy, Focal Brachytherapy , Assessment of QOL

INTERVENTIONS:
Other: Prostate Biopsy, Focal Brachytherapy , Assessment of QOL — A re-staging transrectal or transperineal ultrasound-guided prostate biopsy as currently performed at participating institutions. Focal brachytherapy will be performed at 8 weeks following the transrectal or transperineal biopsy or sooner if the patient has recovered from the repeat biopsy and the treating physician determines it is safe to proceed with treatment. The regions will be targeted with the prescription dose and receive 144 Gy of Iodine-125 (I-125). The quality-of-life assessment will focus on erectile function, urinary function, bowel function, and general health related quality of life. The patients will complete this assessment at baseline and then approximately 3 ± 1 months, 6 ± 1 months, 12 ± 2 months, 18 ± 2 months, and 24 ± 2 months after treatment.

SUMMARY:
The purpose of this study is to see what side effects a type of radiation treatment called focal brachytherapy has in treating early stage prostate cancer. The study is also looking at how useful focal brachytherapy will be in treating prostate cancer. Additionally, the investigators would like to see how this type of treatment impacts quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥ 21 years of age with a life expectancy estimated to be > 10-years.
* Diagnosis of adenocarcinoma of the prostate confirmed by MSKCC or participating site pathology review.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Prostate cancer clinical stage T1c-T2a
* PSA < 10ng/mL (this will be the PSA level prompting the prostate biopsy)
* MRI evidence of one-sided disease performed within 3 months of registration
* Prostate size <60 cc at time of treatment- if the prostate is larger, hormonal therapy is allowed to achieve the required size Screening biopsy parameters:
* Minimum of 10 biopsy cores
* Gleason grade 7 in two cores or less, with no primary Gleason grade 4 or 5 in any cores
* Unilateral cancer (only right-sided or left-sided, not bilateral)
* No more than 50 % cancer in any one biopsy core
* No more than 25 % of cores containing cancer
* Repeat transrectal or transperineal prostate biopsy that must meet the following parameters:
* Minimum of 12 biopsy cores
* Unilateral cancer (only right-sided or left-sided, not bilateral)
* Gleason grade 7 in two cores or less, with no primary Gleason grade 4 or 5 in any cores
* No more than 50 % cancer in any one biopsy core
* No more than 25 % of cores containing cancer

Subject Exclusion Criteria:

* Medically unfit for anesthesia
* Evidence or suspicion of extracapsular extension on MRI
* IPSS score > 18
* Unable to receive MRI
* Prior radiotherapy for the current disease

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-05; Primary Completion 2017-10-06 (Actual); Study Completion 2017-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zelefsky, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - North Shore LIJ, New Hyde Park, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Md Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prostate Biopsy, Focal Brachytherapy , Assessment of QOL
Started | 3
Completed | 1
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Prostate Biopsy, Focal Brachytherapy , Assessment of QOL
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 57 [50 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Late Toxicity Outcomes
Description: focal brachytherapy in patients with low risk prostate cancer This study will utilize the toxicity grading scale Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Time Frame: 6 months to 2 years
Population: Data not collected
Arm/Group | Prostate Biopsy, Focal Brachytherapy , Assessment of QOL
Number analyzed (Participants) | 0

2. Secondary Outcome: To Evaluate the Local Tumor Control After Focal Brachytherapy
Description: as measured by the ability to obtain all negative biopsy cores 12 and 24 months after completion of therapy in the hemi-gland of where the focal therapy was administered. "All negative" means no prostate cancer;
Time Frame: 12 and 24 months
Population: Data not collected
Arm/Group | Prostate Biopsy, Focal Brachytherapy , Assessment of QOL
Number analyzed (Participants) | 0

3. Secondary Outcome: To Evaluate the Change From Baseline in QOL Indicators
Description: Following focal brachytherapy in patients with early stage low volume localized prostate cancer. The scales to measure these domains were derived from the previously validated MSKCC Prostate-Health Related Quality of Life Questionnaire (PHRQOLQ
Time Frame: baseline and then approximately 3 ± 1 months, 6 ± 1 months, 12 ± 2 months, 18 ± 2 months, and 24 ± 2 months after treatment
Population: Data not collected
Arm/Group | Prostate Biopsy, Focal Brachytherapy , Assessment of QOL
Number analyzed (Participants) | 0

4. Secondary Outcome: To Correlate Post-treatment MRI Findings With Post-treatment Biopsy Outcomes
Description: Post-treatment MRI outcome is defined as a 3-level categorical variable: positive, negative and undetermined. Post-treatment biopsy outcome is defined as a binary variable: positive and negative. We will examine the correlation between the 12-month MRI and 12-month biopsy, and between the 24-month MRI and 24-month biopsy. The correlation will be assessed by a Fisher exact test.
Time Frame: 2 years
Population: Data not collected
Arm/Group | Prostate Biopsy, Focal Brachytherapy , Assessment of QOL
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Prostate Biopsy, Focal Brachytherapy , Assessment of QOL
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prostate Biopsy, Focal Brachytherapy , Assessment of QOL (N=3)
Fecal incontinence (Gastrointestinal disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Alanine aminotransferase increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-11-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT01354951/Prot_SAP_000.pdf